CLINICAL TRIAL: NCT00922168
Title: Pre-operative PSG Assessment of Cardiac Surgery Inpatients
Brief Title: Pre-operative Polysomnography Assessment of Cardiac Surgery Inpatients
Status: Completed | Type: Observational
Sponsor: Cleveland Medical Devices Inc (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); The Cleveland Clinic (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: Pre-op PSG; R44NS042451 (NIH)
Record Dates: First submitted 2009-06-15; First posted 2009-06-17 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea; Central Sleep Apnea
Keywords: Sleep; apnea; obstructive; central
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Apnea, Central; Apnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Surgeries: CABG, valve replacements

SUMMARY:
The purpose of this study is to assess the prevalence and morbidity rates of sleep disordered breathing in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing major cardiovascular surgery (coronary artery bypass graft, valve replacement surgery, or aortic surgery) under general anesthesia.
* Subjects in whom surgery is planned for greater than 1 day but less than 60 days from the time of enrollment.

Exclusion Criteria:

* Subjects treated for sleep apnea with positive airway pressure (PAP) therapy or oral appliance in the past 30 days.
* Subjects undergoing Maze procedure for atrial fibrillation.
* Subjects unable to comply with study procedures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cardiac surgery patients
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2007-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of Sleep Disordered Breathing in Cardiac Surgery Patients | September 2009

SECONDARY OUTCOMES:
Assess Post-Operative Complications of Patients with Sleep Disordered Breathing | September 2009

CONTACTS AND LOCATIONS:
Overall Officials: Hani A Kayyali, MS, Principal Investigator — Cleveland Medical Devices Inc; Nancy Foldvary, DO, Principal Investigator — The Cleveland Clinic; Nancy Collop, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Cleveland Clinic Foundation, Cleveland, Ohio